CLINICAL TRIAL: NCT02518867
Title: Modulating and Managing the Motor Disability of Children With Cerebral Palsy Using Motor Transcranial Magnetic Stimulation
Brief Title: Motor Disability of Children With Cerebral Palsy Using Motor Transcranial Magnetic Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98-0118A
Record Dates: First submitted 2015-02-10; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Transcranial magnetic stimulation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- high intensity iTBS (Experimental): high intensity iTBS: 100% of active motor threshold for 3 days.
  Interventions: Other: high intensity iTBS
- low intensity iTBS (Experimental): low intensity iTBS: 80% of active motor threshold for 3 days.
  Interventions: Other: low intensity iTBS
- sham iTBS (Sham Comparator): sham iTBS for 3 days.
  Interventions: Other: sham iTBS

INTERVENTIONS:
Other: high intensity iTBS — In intermittent theta burst stimulation pattern (iTBS) will intermittently give a 2 s train of TBS every 10s for a total of 20 times (high intensity , 100% of active motor threshold) TBS for 3 days.
  Other Names: high intensity intermittent theta burst stimulation
  Arms: high intensity iTBS
Other: low intensity iTBS — In intermittent theta burst stimulation pattern (iTBS) will intermittently give a 2 s train of TBS every 10s for a total of 20 times (low intensity, 80% of active motor threshold) TBS for 3 days.
  Other Names: low intensity intermittent theta burst stimulation
  Arms: low intensity iTBS
Other: sham iTBS — In sham burst stimulation pattern (sham TBS) will intermittently give a sham TBS treatment.
  Other Names: sham theta burst stimulation
  Arms: sham iTBS

SUMMARY:
Transcranial magnetic stimulation (TMS) has opened new potential avenues for the treatment of neuropsychiatric diseases via the effects of modulation on neuroplasticity. Repetitive TMS (rTMS) is a non-invasive method of stimulation neural pathways in the brain of conscious subjects through the intact scalp. The investigators hypothesize that excitatory rTMS applied over the motor cortex would increase motor cortex activity and result in an increase in the inhibitory input through the corticospinal tract to the spinal cord, thus reducing alpha neuron hyperactivity and consequently clinical spasticity. In this study, the investigators will apply the stimulation on the legs motor cortex area, which can cover supplemental motor area (SMA). Therefore, not only the spasticity, but also the motor control of legs both can be modulated by stimulation. Theta burst stimulation is a condition of rTMS which was designed by the co-investigator. It has controllable, consistent, long-lasting, and powerful effects on motor cortex physiology and behavior. The investigators therefore design this protocol using theta burst stimulation on the motor cortex of the patients of cerebral palsy. The investigators expect that there would be an effect on the reduction of spasticity after rTMS on the brain of children with CP, thus improving the motor control of legs.

DETAILED DESCRIPTION:
In this study, the investigators design 3 steps to find out the optimal condition of rTMS for the treatment and managing of motor disability of CP. The first is to find out the optimal intensity of rTMS. The second is to find out the optimal duration of rTMS and long term effects. The third is to compare the effectiveness of botulinum toxin injection, rTMS, and combined therapy (botulinum toxin injection and rTMS) for children with CP.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild to moderate CP with spastic diplegia or hemiplegia according to clinical criteria
* age 7-20 years
* no use of botulinum toxin in the past 4 months
* no significant perceptual or communication disturbances
* no other peripheral or central nervous system dysfunction
* no active inflammatory or pathologic changes in lower limb joints during the previous 6 months
* no active medical problems, such as pneumonia, upper gastrointestinal bleeding, or urinary tract infection
* no active problems of epilepsy and EEG without epileptiform discharge
* ability to walk 20m without walking aids, such as a cane, quadricane or walker

Exclusion Criteria:

* Metabolic disorders, such as inborn error of metabolism, electrolyte, and endocrine disorders.
* Active infectious disease, such as meningitis and encephalitis.
* Patients with active medical problems, such as pneumonia, upper gastrointestinal bleeding, or urinary tract infection.
* Poor compliance or intolerance for the TMS therapy
* Subjects with metallic implants or pregnancy.
* EEG show epileptiform discharge

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Kinematic analysis in post-treatment (after 3 days intervention) and one months follow up. | baseline, post-treatment (after 3 days intervention), one months
  Kinematic analysis for gait analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Lin Lin, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan